CLINICAL TRIAL: NCT02299349
Title: Bupivacaine Liposome Suspension Versus a Concentrated Multi Drug Periarticular Injection in 70 Patients Undergoing Total Knee Arthroplasty Without Femoral Nerve Block: a Double-blinded, Randomized Clinical Trial
Brief Title: Bupivacaine Liposome Suspension Versus a Concentrated Multi Drug Periarticular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13055-13-034
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2017-03

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine liposome suspension (Experimental): bupivacaine liposome suspension periarticular injection
  Interventions: Drug: bupivacaine liposome suspension
- concentrated multi drug injection (Active Comparator): concentrated multi drug periarticular injection
  Interventions: Drug: concentrated multi drug Ketorlac, Morphine PF, Epinephrine, Ropivicaine, 0.9% NaCL

INTERVENTIONS:
Drug: bupivacaine liposome suspension — bupivacaine liposome suspension periarticular injection
  Other Names: Exparel
  Arms: bupivacaine liposome suspension
Drug: concentrated multi drug Ketorlac, Morphine PF, Epinephrine, Ropivicaine, 0.9% NaCL — Ketorolac 30 mg, Morphine PF 5 mg, Epinephrine 0.6 mg, Ropivacaine 400 mg, QS to 100ml with 0.9% NaCl
  Other Names: Ketorlac, Morphine PF, Epinephrine, Ropivicaine, 0.9% NaCL
  Arms: concentrated multi drug injection

SUMMARY:
Despite a robust multimodal pain management regimen, patients undergoing total knee arthroplasty (TKA) continue to report low satisfaction with postoperative pain management. Patient satisfaction further declines with any adverse event such as a drug reaction to neuroleptic medications or a patient fall due to a femoral nerve block. A new method of pain management throughout the hospital experience is warranted to improve patient satisfaction and the possibility of related adverse events. The purpose of this study is to examine if there is a difference in post operative pain and morphine (MSO4) total consumption for hospitalized TKA patients without femoral nerve block receiving an intra-operative periarticular injection of bupivacaine liposome suspension versus a concentrated multi drug.

DETAILED DESCRIPTION:
The void in the literature is that while multimodal pain management reduces postoperative pain in the majority of TKA patients6-14, too many are still dissatisfied with overall pain control13 and adverse drug reactions (dizziness and somnolence) to neuroleptic medications15. Additionally, postoperative falls are greater with femoral nerve blocks16, and new neurological symptoms are associated with the block17. Bupivacaine liposome suspension periarticular injection has large scale national anecdotal support for TKA pain control with avoidance of regional block adversity. There is one recent randomized control trial in TKA patients favorably comparing periarticular injection with bupivacaine liposome suspension versus bupivacaine hydrochloride (HCL)5. To date the clinical use and published evidence most robustly supports bupivacaine liposome suspension in patients undergoing bunionectomy or hemorrhoidectomy. Additionally, in preparation for shorter hospital stays for total joint arthroplasty, a more effective and better tolerated pain management solution is needed.

Hypothesis Statement:

Hospitalized TKA patients without a pre-operative femoral nerve block will experience improved postoperative pain control and less MSO4 equivalence consumption when receiving an injection of bupivacaine liposome suspension versus concentrated multi drug.

ELIGIBILITY:
Inclusion Criteria:

* TKA candidacy
* Osteoarthritis
* Failure of non-operative treatments to control knee pain
* Patients able to understand and agree to study inclusion

Exclusion Criteria:

* Subjects have orthopaedic and medical co-morbidities that would thwart postoperative pain control such as extra-articular pathology with referred pain to the knee (spinal stenosis, neuropathy,ipsilateral hip disease)
* Severe knee deformity
* Post-traumatic and inflammatory arthritis
* BMI above 40
* Patients unable to receive multimodal pain remitting agents
* Active knee sepsis
* Remote sites of active infection
* Diabetes with A1C > 7
* ASA class > lll
* Cardiac disease failing medical clearance
* Severe liver disease
* PAD with AAI < 0.75
* Seizure disorder
* Allergic to any pain remitting agent
* Alcohol abuse
* Smoking abuse

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine Liposome Suspension | Concentrated Multi Drug Injection
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Men and women aged 18 and up receiving total knee arthroplasty for degenerative joint disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Liposome Suspension | Concentrated Multi Drug Injection | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.3) | 65.6 (7.9) | 66.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 22 | 15 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 35 | 34 | 69
  African American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores (Visual Analog Pain Scores)
Description: visual analog pain scores (scale 0=no pain; 10=worst pain imaginable)
Time Frame: 1 day following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine Liposome Suspension | Concentrated Multi Drug Injection
Number analyzed (Participants) | 35 | 35
units on a scale | 2.6 (1.27) | 3.3 (1.55)

2. Secondary Outcome: MS04 Equivalent Consumption
Description: in hospital total MS04 equivalent consumption
Time Frame: 1 day following surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Bupivacaine Liposome Suspension | Concentrated Multi Drug Injection
Number analyzed (Participants) | 35 | 35
mg | 10.0 [5.0 to 15.0] | 15.0 [8.0 to 20.0]

ADVERSE EVENTS:
Arm/Group | Bupivacaine Liposome Suspension | Concentrated Multi Drug Injection
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes